CLINICAL TRIAL: NCT07344636
Title: Temporal and Dose-response Effects of Nicotinamide Riboside Supplementation on Metabolic Flexibility During Zone 2 Training in Adults: a Double-blinded, Randomized, Controlled, Crossover Trial
Brief Title: Effects of NR Supplementation on Metabolic Flexibility in Zone 2 Training
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ZHANG Jiaqi (Other)
Responsible Party: Sponsor-Investigator, ZHANG Jiaqi, Principal Investigator, Chinese University of Hong Kong
Organization: Chinese University of Hong Kong (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: SBRE-25-0349
Record Dates: First submitted 2026-01-05; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Health Adult Subjects
MeSH Terms: interventions — nicotinamide-beta-riboside

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 600 mg (Experimental)
  Interventions: Dietary Supplement: Nicotinamide Riboside (NR)
- 300 mg (Experimental)
  Interventions: Dietary Supplement: Nicotinamide Riboside (NR)
- 0 mg (No Intervention)

INTERVENTIONS:
Dietary Supplement: Nicotinamide Riboside (NR) — 600 mg NR
  Arms: 600 mg
Dietary Supplement: Nicotinamide Riboside (NR) — 300 mg NR
  Arms: 300 mg

SUMMARY:
Zone 2 training, a low-intensity endurance exercise performed at approximately 66-80% of VO₂max or near the first ventilatory threshold, has gained popularity for improving aerobic capacity, fat metabolism, and mitochondrial efficiency. It preserves glycogen stores and delays fatigue, making it an essential training method for both athletes and recreational exercisers. Nicotinamide adenine dinucleotide (NAD) is a vital metabolite that regulates cellular energy metabolism and redox homeostasis. It participates in oxidative reactions within the tricarboxylic acid cycle and electron transport chain, sustaining ATP synthesis and mitochondrial efficiency. Exercise influences multiple pathways of NAD metabolism, altering the NAD⁺/NADH ratio and thereby affecting energy production and fatigue resistance. Studies have shown that both aerobic exercise and NAD precursor supplementation (e.g., nicotinamide riboside [NR]) can elevate body NAD levels and enhance mitochondrial function, though findings remain inconsistent due to variations in dosage and participants' characteristics. This study aims to investigate how acute NR supplementation interacts with Zone 2 cycling training in adults. Specifically, it examines the temporal and dose-dependent effects of NR supplementation on metabolic flexibility and exercise performance. The results may clarify the potential synergistic benefits of combining NAD supplementation with low-intensity endurance training to improve aerobic adaptability.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old
* BMI <30 kg/m2

Exclusion Criteria:

* Present of health conditions that contraindicate participation in exercise training, such as a history of cardiovascular disease, cancer, or musculoskeletal disorders
* Currently taking vitamin B supplements and/or NAD precursors
* Taking medication that may affect the test results

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Substrate utilization (CHO and fat oxidation rate) | From enrollment to the end of treatment at 4 weeks

SECONDARY OUTCOMES:
Oxygen consumption | From enrollment to the end of treatment at 4 weeks
Heart rate | From enrollment to the end of treatment at 4 weeks
Blood glucose concentration | From enrollment to the end of treatment at 4 weeks
Blood lactate concentration | From enrollment to the end of treatment at 4 weeks
Peak power output | From enrollment to the end of treatment at 4 weeks
Mean power output | From enrollment to the end of treatment at 4 weeks
Rating of perceived exertion | From enrollment to the end of treatment at 4 weeks
Muscle pain scale | From enrollment to the end of treatment at 4 weeks
  Muscle pain scale is a 5-point likert scale ranging from "1- Not at all" to "5- Extreme", with higher value indicating muscle pain.
Muscle fatigue scale | From enrollment to the end of treatment at 4 weeks
  Muscle fatigue scale is a 5-point likert scale ranging from "1- Not at all" to "5- Extreme", with higher value indicating muscle fatigue.

OTHER OUTCOMES:
Height | From enrollment to the end of treatment at 4 weeks
Weight | From enrollment to the end of treatment at 4 weeks
Power output at VT1 | From enrollment to the end of treatment at 4 weeks
Health history questionnaire | From enrollment to the end of treatment at 4 weeks
  This questionnaire includes questions regarding participant's present/past history of diseases and his/her family history of diseases.
International Physical Activity Questionnaire (IPAQ) | From enrollment to the end of treatment at 4 weeks
  IPAQ is a validated questionnaire to measure the physical activity of participants during the past 7 days. The score will be transformed to metabolic equivalents of tasks per week (METs/week), with higher value indicating greater participation in physical activity.

IPD SHARING:
Plan to Share IPD: Undecided